CLINICAL TRIAL: NCT02835768
Title: Effectiveness of Internet-based Injury Prevention Program in Enhancing Mother's Knowledge on Child Safety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: injury prevention; 08150345 (Other Grant/Funding Number: Health Care and Promotion Fund of the Food and Health Bureau, the Hong Kong Government)
Record Dates: First submitted 2016-06-13; First posted 2016-07-18 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Child Safety; Injury Prevention; Internet-based Intervention; Anticipatory Guidance; Chinese Mothers

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Outcomes Assessor

ARMS (2):
- Intervention (Experimental): Each participant will be provided an information package - the parenting booklet from Maternal and Child Health Centres (MCHCs) about domestic safety tips. Participants will be given an additional leaflet about the domestic safety website with address link and brief introductory information.
  Interventions: Other: Internet-based injury prevention program
- Control (No Intervention): Each participant will be provided an information package - the parenting booklet from Maternal and Child Health Centres (MCHCs) about domestic safety tips. Only this booklet serves as the anticipatory guidance to mothers about domestic safety.

INTERVENTIONS:
Other: Internet-based injury prevention program — An injury prevention website serves as the Internet-based intervention providing two key topics: 1) Types of domestic injury, and 2) how to prevent different types of domestic injury. The domestic injury prevention information "Home Safety Tips" is divided into four subgroups according to various safety issues relevant to infants/children's age groups. Apart from a knowledge hub, the website incorporates additional functions of feedback counselling, video demonstration, online consultation, games, safety checklist and discussion forum.
  Arms: Intervention

SUMMARY:
Background: Provision of anticipatory guidance to parents is recommended as an effective strategy to prevent injuries among young children. Internet-based anticipatory guidance is suggested to reinforce the effectiveness of injury prevention, and improve parents' knowledge on child safety. Parents receiving the guidance can reduce children's exposure to injury risk by adopting better childcare practices and using appropriate child safety devices at home.

Objective: This study will examine the effectiveness of Internet-based injury prevention program with parental anticipatory guidance in enhancing mothers' knowledge on child safety. It aims at increasing mothers' knowledge and motivation of learning about domestic injury prevention through a new Internet-based intervention model. It also targets to improve mothers' attitude and perceived behavioral control of domestic safety practice.

Methods: The study would adopt a randomized controlled trial design and recruit 934 mothers from the antenatal clinics and postnatal wards of two major public hospitals in Hong Kong. Participating mothers will be randomized into the intervention or control group with equal likelihood. Mothers in intervention group will be provided with free access to an Internet-based injury prevention program with anticipatory guideline whereas those in the control group will receive relevant parenting booklet.

Results: It is hypothesized that mothers' general and age-appropriate knowledge on child safety and motivation of learning about domestic injury prevention as the primary outcome measures will be enhanced.

Conclusions: The Internet is increasingly recognized as a practical and cost-effective platform for health education and safety information delivery. The goals of this study are to examine the effectiveness of a new Internet-based intervention program for improving mothers' knowledge, and raising mothers' awareness about the importance and consequences caused by domestic injuries.

ELIGIBILITY:
Inclusion Criteria:

* Mothers attending the antenatal clinics/staying in the postnatal wards at Kwong Wah Hospital or Queen Mary Hospital.

Exclusion Criteria:

* Mothers unable to read Chinese and those without access to Internet.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1012 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change of general safety knowledge | At the beginning of the study and infants' ages of 18-month-old
  This component aims to evaluate mothers' general knowledge change related to domestic injury prevention. Questions will be designed as statement format and two key topics will be covered in the questionnaire: common childhood domestic injuries and safety precautions
2-month-old safety knowledge | At infants' ages of 2-month-old
  This component examines 2-month-old domestic safety related knowledge, intention, attitude and perceived behavioral control of safety practice. The questionnaire consists of multiple-choice questions. This quiz answering design targeted to reinforce safety concepts as well as to sustain knowledge enhancement.
6-month-old safety knowledge | At infants' ages of 6-month-old
  This component examines 6-month-old domestic safety related knowledge, intention, attitude and perceived behavioral control of safety practice. The questionnaire consists of multiple-choice questions. This quiz answering design targeted to reinforce safety concepts as well as to sustain knowledge enhancement.
9-month-old safety knowledge | At infants' ages of 9-month-old
  This component examines 9-month-old domestic safety related knowledge, intention, attitude and perceived behavioral control of safety practice. The questionnaire consists of multiple-choice questions. This quiz answering design targeted to reinforce safety concepts as well as to sustain knowledge enhancement.
12-month-old safety knowledge | At infants' ages of 12-month-old
  This component examines 12-month-old domestic safety related knowledge, intention, attitude and perceived behavioral control of safety practice. The questionnaire consists of multiple-choice questions. This quiz answering design targeted to reinforce safety concepts as well as to sustain knowledge enhancement.
18-month-old safety knowledge | At infants' ages of 18-month-old
  This component examines 18-month-old domestic safety related knowledge, intention, attitude and perceived behavioral control of safety practice. The questionnaire consists of multiple-choice questions. This quiz answering design targeted to reinforce safety concepts as well as to sustain knowledge enhancement.

SECONDARY OUTCOMES:
Website usage statistics | 18 months
  Participants will be required to register as a member in order to assess the website. The investigators will be able to record all the actions taken by each user.
Website user acceptance | At the end of the study, an average of 18 months
  Towards the end of the intervention period, subjects will be reminded to complete a modified user acceptance evaluation from IBM Computer Usability Satisfaction Questionnaires. The practicability of the Internet-based domestic injury prevention website will be evaluated in terms of its layout, structure, usability, readability, accessibility and ease of navigation.

REFERENCES:
- [Derived] Chow CB, Wong WH, Leung WC, Tang MH, Chan KL, Or CK, Li TM, Ho FK, Lo D, Ip P. Effectiveness of a Technology-Based Injury Prevention Program for Enhancing Mothers' Knowledge of Child Safety: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2016 Oct 31;5(4):e205. doi: 10.2196/resprot.6216. PMID 27799138